CLINICAL TRIAL: NCT04243148
Title: Frailty in Patients With Cirrhosis: Prognostic Value of the Phase Angle in Hospitalized Patients and Effect of a Multifactorial Intervention (Home Exercise, Branched-chain Aminoacids and Probiotic)
Brief Title: Frailty in Patients With Cirrhosis: Prognostic Value of the Phase Angle in Hospitalized Patients and Effect of Multifactorial Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-FRA-2019-36
Record Dates: First submitted 2020-01-14; First posted 2020-01-28 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-07

CONDITIONS: Cirrhosis of the Liver; Sarcopenia; Frailty Syndrome
Keywords: Falls; Hospitalizations; Mortality; Phase angle; Body Composition
MeSH Terms: conditions — Fibrosis; Sarcopenia; Frailty | interventions — Amino Acids, Branched-Chain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multifactorial intervention (Experimental): Frail and pre-frail patients will receive multifactorial intervention consisting of home exercise, BCAA supplements and a multispecies probiotic for 12 months.
  Interventions: Combination Product: Home exercise program for 12 months.; Combination Product: Multispecies probiotic: Vivomixx®; Combination Product: Branched-chain amino acids (BCAA)
- Control group (Experimental): Frail and pre-frail patients will be followed but will not receive any specific intervention.
  Interventions: Combination Product: No specific intervention.

INTERVENTIONS:
Combination Product: Home exercise program for 12 months. — Physical exercise at home: At the beginning of the study, group sessions will be conducted with 5 patients of 1-hour duration, where they will be taught the individualized program according to their physical condition and they will be given the necessary material (pedaling, dumbbells and elastic bands) and paper support on the program, also using the Vivifrail method through infographics. The group session will be repeated every 3 months to check the compliance of the program by reviewing daily activity, evaluate possible problems and review the exercises. The program will consist of aerobic and anaerobic exercise by pedaling (cardiovascular resistance) and resistance exercises with dumbbells and elastic bands (muscular strength), flexibility training by stretching, and coordination and balance exercises. Patients will perform 3 sessions per week of 20-30 min. increasing progressively according to tolerance up to 45-60 min. each.
  Arms: Multifactorial intervention
Combination Product: Multispecies probiotic: Vivomixx® — Multispecies probiotic: Vivomixx® is a probiotic mixture of 8 bacterial strains:
  Streptococcus thermophilus DSM 24731® / NCIMB 30438, Bifidobacterium breve DSM 24732® / NCIMB 30441, Bifidobacterium longum DSM 24736® / NCIMB 30435*, Bifidobacterium infantis DSM 24737® / NCIMB 30436*, Lactobacillus acidophilus DSM 24735® / NCIMB 30442, Lactobacillus plantarum DSM 24730® / NCIMB 30437, Lactobacillus paracasei DSM 24733® / NCIMB 30439, Lactobacillus delbrueckii subsp. bulgaricus DSM 24734® / NCIMB 30440**
  * Re-classified as B. lactis ** Re-classified as L. helveticus The active agent will be supplied as an envelope of 4.4 g with a dose of 450x109 million live bacteria per envelope with maltose and silicon dioxide as excipients, administered 2 times/day throughout the study.
  Arms: Multifactorial intervention
Combination Product: Branched-chain amino acids (BCAA) — Branched-chain amino acids (BCAA): In addition to the exercise program and the probiotic, patients in the intervention group will receive BCAA supplements (powder in 8:1:1 ratio in favor of L-leucine) 10 g 30-60 min. before the exercise session throughout the study, in order to enhance the effect of exercise on muscle mass and improve cognitive function. We have chosen this dose based on the literature data and the satisfactory results obtained with this dose in our previous study. BCAA supplements will be supplied by the Pharmacy Service of our center.
  Arms: Multifactorial intervention
Combination Product: No specific intervention. — Follow up as a clinical practice
  Arms: Control group

SUMMARY:
This study evaluate Frailty syndrome (FS) as a common syndrome in patients with cirrhosis and it is an independent predictor of hospitalizations, falls and mortality. Identifying, treating and preventing FS can improve the prognosis and quality of life of these patients and reduce health costs.

DETAILED DESCRIPTION:
Substudy I. The phase angle (PA) determined by electrical bioimpedance is an index of FS with prognostic value in outpatients with cirrhosis, but its usefulness in hospitalized patients has not been studied. Objective: To analyze the prognostic value of PA in hospitalized patients with cirrhosis. Patients and Methods: 100 hospitalized patients with cirrhosis will be consecutively included and PA will be determined by bioimpedance at admission. The correlation between PA and liver function and frailty markers, and the evolution during hospitalization, as well as the incidence of falls, hospitalizations and mortality during follow-up will be analyzed. Substudy II. Given the multidimensional nature of the FS, we propose a multifactorial non-pharmacological intervention based on evidence from previous studies that could be implemented in daily clinical practice. Objective: To evaluate if a multifactorial intervention can improve the FS and decrease the related events (hospitalizations, falls and mortality) in patients with cirrhosis. Patients and Methods: 150 outpatients with cirrhosis will be included and evaluated using the Liver Frailty Index. Frail and pre-frail patients will be randomized into two groups: one group that will receive a multifactorial intervention, consisting of exercise at home, branched-chain amino acids and multispecies probiotic for one year, and one control group. The evolution of the Liver Frailty Index and other parameters (muscle and cognitive function, bioimpedance, risk of falls, quality of life) and biomarkers (miostatin, immune response, microbiota) of FS, and the incidence of hospitalizations, falls and mortality in both groups will be prospectively analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Aged >18 years old, with cirrhosis diagnosed by clinical, analytical and ultrasound criteria or liver biopsy
* Conscious and oriented in time and space and able to understand and follow the indications of the study.

Exclusion Criteria:

* Liver cirrhosis with poor prognosis (MELD [Model for End Stage Liver Disease]> 25)
* Hepatocellular carcinoma or other active neoplastic disease
* Expected survival <6 months
* Acute and/or chronic hepatic encephalopathy
* Neurological disorder that hinders the performance of the tests
* Active alcoholism in the previous 3 months
* Severe comorbidities
* Hospitalization in the previous month
* Contraindications to exercise or probiotic treatment (immunosuppression)
* Refusal to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Substudy I: Mortality during hospitalization and follow-up | One year
  At the time of admission, during hospitalization and in one hundred outpatients visits every 3 months until 12 months of follow-up
Substudy II: Evolution of the Liver Frailty Index. | One year
  At the beginning and every 3 months in one hundred fifty outpatient visits until the end of the study at 12 months

SECONDARY OUTCOMES:
Phase angle (PA) | One year
  By bioimpedance (BIA 101 with Bodygram Pro software, Akern) at admission, hospital discharge and every 3 months.
Degree of sarcopenia | One year
  Grip strength assessed by a dynamometer (KERN MAP 80K1, Akern). The results will be adjusted by age and gender
Biomarkers of frailty | One year
  At baseline and at 12 months.We will quantify by specific ELISA kits and multiplex assays biomarkers
Fall risk tests | One year
  Walking speed (41) and Timed Up & Go: time in seconds that the patient uses to get up from a chair, walk 3 meters and sit back without support. Times greater than 9 seconds to travel the distance is considered a risk of falls
Cognitive function | One year
  Psychometric Hepatic Encephalopathy Score (PHES). Scores <-4 points is considered as a cognitiva impairment
Degree of Quality of life | One year
  SF-36 questionnaire
  - Scores above 50 will be better and below 50 points will be worse.
Fecal microbiota | One year
  At baseline, 6 and 12 months.For the extraction of genomic DNA from stool samples, a previous protocol according to the International consortium (IHMS: http://www.microbiome-standards.org/) will be used.
Degree Quality of life | One year
  Depression and anxiety scale (HADS): Scores higher than 11 are probably cases in each of the subscales

CONTACTS AND LOCATIONS:
Overall Officials: Germán Soriano, PhD, Principal Investigator — Hospital Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vega-Abellaneda S, Roman E, Soler Z, Ortiz MA, Rossi G, Biagini L, Sanchez E, Pons-Tarin M, Laghi L, Mengucci C, Kaur N, Poca M, Cuyas B, Serrano-Gomez G, Alvarado E, Manichanh C, Soriano G. A Metagenomics Approach to Frailty in Patients With Cirrhosis Undergoing a Multifactorial Intervention. Liver Int. 2025 Dec;45(12):e70418. doi: 10.1111/liv.70418. PMID 41174950
- [Derived] Roman E, Kaur N, Sanchez E, Poca M, Padros J, Nadal MJ, Cuyas B, Alvarado E, Vidal S, Ortiz MA, Hernandez E, Santesmases R, Urgell E, Juanes E, Ferrero-Gregori A, Escorsell A, Guarner C, Soriano G. Home exercise, branched-chain amino acids, and probiotics improve frailty in cirrhosis: A randomized clinical trial. Hepatol Commun. 2024 May 3;8(5):e0443. doi: 10.1097/HC9.0000000000000443. eCollection 2024 May 1. PMID 38701490